CLINICAL TRIAL: NCT05059262
Title: A Phase 3, Randomized, Placebo-controlled, Double-blind Study of Vimseltinib to Assess the Efficacy and Safety in Patients With Tenosynovial Giant Cell Tumor (MOTION)
Brief Title: Study of Vimseltinib for Tenosynovial Giant Cell Tumor
Acronym: MOTION
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCC-3014-03-001; 2024-513624-42-00 (EU CTIS Number)
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Results first posted 2025-02-24 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Tenosynovial Giant Cell Tumor; Pigmented Villonodular Synovitis; Giant Cell Tumor of Tendon Sheath; Tenosynovial Giant Cell Tumor, Diffuse; Tenosynovial Giant Cell Tumor, Localized
Keywords: TGCT; PVNS
MeSH Terms: conditions — Giant Cell Tumor of Tendon Sheath; Synovitis, Pigmented Villonodular

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1/Part 2 - Vimseltinib/Vimseltinib (Experimental): Participants received blinded treatment of 30 mg twice a week (BIW) vimseltinib for 24 weeks in Part 1 and open-label 30 mg BIW vimseltinib in Part 2.
  Interventions: Drug: Vimseltinib
- Part 1/Part 2: Placebo/Vimseltinib (Placebo Comparator): Participants received blinded treatment of BIW matching placebo for 24 weeks in Part 1 and open-label 30 mg BIW vimseltinib in Part 2.
  Interventions: Drug: Vimseltinib; Drug: Placebo

INTERVENTIONS:
Drug: Vimseltinib — Administered orally
  Other Names: DCC-3014
Drug: Placebo — Administered orally
  Arms: Part 1/Part 2: Placebo/Vimseltinib

SUMMARY:
This is a multicenter Phase 3 clinical study, which aims to evaluate the effectiveness of an investigational drug called vimseltinib for the treatment of tenosynovial giant cell tumor (TGCT) in cases where surgical removal of the tumor is not an option.

The study consists of two parts. In Part 1, eligible study participants will be assigned to receive either vimseltinib or matching placebo for 24 weeks. A number of assessments will be carried out during the course of the study, including physical examinations, blood tests, imaging studies, electrocardiograms, and questionnaires. MRI scans will be used to evaluate the response of the tumors to the treatment. Participants assigned to placebo in Part 1 will have the option to receive vimseltinib for Part 2. Part 2 is a long-term treatment phase in which all participants receive open-label vimseltinib.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age
2. TGCT for which surgical resection is not an option (tumor biopsy to confirm diagnosis required if no histology/pathology available at screening)
3. Symptomatic disease as defined as at least moderate pain or at least moderate stiffness (defined as a score of 4 or more, with 10 describing the worst condition) within the screening period and documented in the medical record
4. Participants should complete 14 consecutive days of questionnaires during the screening period and must meet minimum requirements as outlined in study protocol
5. Must have stable analgesic regimen, as judged by the investigator, for at least 2 weeks prior to first dose of study drug
6. Must have measurable disease, as per RECIST Version 1.1, with at least one lesion having a minimum size of 2cm
7. Adequate organ and bone marrow function
8. If a female of childbearing potential, must have a negative pregnancy test prior to enrollment and agree to follow the contraception requirements
9. Must provide signed consent to participate in the study and is willing to comply with study-specific procedures
10. Willing and able to complete the patient-reported outcome (PRO) assessments on an electronic device

Exclusion Criteria:

1. Previous use of systemic therapy (investigational or approved) targeting colony-stimulating factor 1 (CSF1) or colony-stimulating factor 1 receptor (CSF1R); previous therapy with imatinib and nilotinib is allowed
2. Received therapy for TGCT, including investigational therapy during the screening period. Participated in a non-TGCT investigational drug study within 30 days of screening.
3. Known metastatic TGCT or other active cancer that requires concurrent treatment (exceptions will be considered on a case-by-case basis)
4. QT interval corrected by Fridericia's formula (QTcF) >450 ms in males or >470 ms in females or history of long QT syndrome
5. Concurrent treatment with any study-prohibited medications
6. Major surgery within 14 days of the first dose of study drug
7. Any clinically significant comorbidities
8. Active liver or biliary disease including nonalcoholic steatohepatitis (NASH) or cirrhosis
9. Malabsorption syndrome or other illness that could affect oral absorption
10. Known active human immunodeficiency virus (HIV), acute or chronic hepatitis B, acute or chronic hepatitis C, or known active mycobacterium tuberculosis infection
11. If female, the participant is pregnant or breastfeeding
12. Known allergy or hypersensitivity to any component of the study drug
13. Contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2021-10-14 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2026-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (35):
- United States (11):
  - City of Hope, Duarte, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - University of Colorado, Aurora, Colorado
  - University of Kansas, Kansas City, Kansas
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Duke Sarcoma Research, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Seattle Cancer Care Alliance, Seattle, Washington
- Chris O'Brien Lifehouse, Camperdown, Australia
- Canada (2):
  - McGill University, Montreal
  - Princess Margaret Hospital, Toronto
- France (3):
  - Institut Bergonié, Bordeaux
  - Centre Léon Bérard, Lyon
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Helios Klinikum Berlin-Buch, Berlin
  - University Hospital Essen (Universitätsklinikum Essen), Essen
- Prince of Wales Hospital, Hong Kong, Hong Kong
- Italy (5):
  - Istituto Ortopedico Rizzoli, Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale", Naples
  - Istituto Oncologico Veneto, Padua
  - Istituto Nazionale Tumori Regina Elena, Rome
- Leiden University Medical Center, Leiden, Netherlands
- Oslo University Hospital, Oslo, Norway
- Klinika Nowotworów Tkanek Miękkich, Kości i Czerniaków Narodowy Instytut Onkologii im. Marii Skłodowskiej-Curie - Państwowy Instytut Badawczy, Warsaw, Poland
- Spain (4):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico San Carlos, Madrid
- Universitäts-Kinderspital beider Basel (UKBB), Basel, Switzerland
- United Kingdom (2):
  - Cancer & Haematology Centre, The Churchill Hospital - Oxford University Hospitals NHS Foundation Trust, London
  - University College London Hospitals, London

REFERENCES:
- [Derived] Gelderblom H, Bhadri V, Stacchiotti S, Bauer S, Wagner AJ, van de Sande M, Bernthal NM, Lopez Pousa A, Razak AA, Italiano A, Ahmed M, Le Cesne A, Tinoco G, Boye K, Martin-Broto J, Palmerini E, Tafuto S, Pratap S, Powers BC, Reichardt P, Casado Herraez A, Rutkowski P, Tait C, Zarins F, Harrow B, Sharma MG, Ruiz-Soto R, Sherman ML, Blay JY, Tap WD; MOTION investigators. Vimseltinib versus placebo for tenosynovial giant cell tumour (MOTION): a multicentre, randomised, double-blind, placebo-controlled, phase 3 trial. Lancet. 2024 Jun 22;403(10445):2709-2719. doi: 10.1016/S0140-6736(24)00885-7. Epub 2024 Jun 3. PMID 38843860
- [Derived] Tap WD, Sharma MG, Vallee M, Smith BD, Sherman ML, Ruiz-Soto R, de Sande MV, Randall RL, Bernthal NM, Gelderblom H. The MOTION study: a randomized, phase III study of vimseltinib for the treatment of tenosynovial giant cell tumor. Future Oncol. 2024 Mar;20(10):593-601. doi: 10.2217/fon-2023-0238. Epub 2023 Aug 18. PMID 37593881

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Presented here is data from the Week 25 primary endpoint analysis. The study is ongoing.
Groups:
- Part 1/Part 2: Vimseltinib/Vimseltinib: Participants received blinded treatment of vimseltinib 30 milligrams (mg) twice a week (BIW) for 24 weeks in Part 1 and open-label vimseltinib 30 mg BIW in Part 2 until end of treatment (EoT).
- Part 1/Part 2: Placebo/Vimseltinib: Participants received blinded treatment of matching placebo BIW for 24 weeks in Part 1 and open-label vimseltinib 30 mg BIW in Part 2 until EoT.
Period: Part 1: Double Blind (Weeks 1 - 24)
Arm/Group | Part 1/Part 2: Vimseltinib/Vimseltinib | Part 1/Part 2: Placebo/Vimseltinib
Started | 83 | 40
Received at Least 1 Dose of Study Drug | 83 | 39
Completed (One participant was continuing in Part 1 of study at time of primary endpoint analysis.) | 75 | 35
Not Completed | 8 | 5
Not completed — Subsequent TGCT therapy and/or surgery | 3 | 0
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Physician Decision | 1 | 1
Not completed — Other reasons | 0 | 1
Not completed — Ongoing in study | 1 | 0
Period: Part 2: Open Label (Weeks 25 - EoS)
Arm/Group | Part 1/Part 2: Vimseltinib/Vimseltinib | Part 1/Part 2: Placebo/Vimseltinib
Started | 74 | 35
Received at Least 1 Dose of Study Drug | 72 | 35
Completed | 0 | 0
Not Completed | 74 | 35
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Ongoing in study | 73 | 32

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Set consisted of participants who were randomized to a study treatment regimen. Presented here are data from Part 1 baseline period.
Groups:
- Part 1/Part 2: Vimseltinib/Vimseltinib: Participants received blinded treatment of vimseltinib 30 mg BIW for 24 weeks in Part 1 and open-label vimseltinib 30 mg BIW in Part 2 until EoT.
- Part 1/Part 2: Placebo/Vimseltinib: Participants received blinded treatment of matching placebo BIW for 24 weeks in Part 1 and open-label vimseltinib 30 mg BIW in Part 2 until end of EoT.
- Total: Total of all reporting groups
Arm/Group | Part 1/Part 2: Vimseltinib/Vimseltinib | Part 1/Part 2: Placebo/Vimseltinib | Total
Number analyzed (Participants) | 83 | 40 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (13.92) | 42.5 (13.67) | 43.4 (13.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 27 | 73
  Male | 37 | 13 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 62 | 23 | 85
  Unknown or Not Reported | 18 | 16 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 0 | 4
  White | 59 | 21 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 19 | 15 | 34

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) at Week 25 Per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1
Description: ORR was assessed by blinded independent radiologic review (IRR) using RECIST Version 1.1. ORR was defined as the percentage of participants who achieved either complete response (CR) or partial response (PR).
  * CR: Disappearance of all target lesions. Any pathological lymph nodes must be <10 millimeter (mm) in short axis. Non-nodal targets must be absent.
  * PR: At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline to Week 25 (Cycle 7, Day 1)
Population: The ITT Set consisted of participants who were randomized to a study treatment regimen.
Measure: Number (95% Confidence Interval); unit: percentage of participants with CR or PR
Groups:
- Vimseltinib: Participants received 30 mg BIW vimseltinib for 24 weeks.
- Placebo: Participants received matching placebo BIW for 24 weeks.
Arm/Group | Vimseltinib | Placebo
Number analyzed (Participants) | 83 | 40
percentage of participants with CR or PR | 39.8 [29.2 to 51.1] | 0 [0.0 to 8.8]
Statistical Analysis 1: Comparison: Vimseltinib vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Stratified by tumor location (lower limb/all other) and region (U.S./non-U.S.) based on Interactive Response Technology (IRT); Difference in ORR = 39.0, 95% CI 2-sided [28.4 to 49.6] — Stratified Mantel-Haenszel with stratification factors based on IRT

2. Secondary Outcome: ORR at Week 25 Per Tumor Volume Score (TVS)
Description: TVS is a semi-quantitative magnetic resonance imaging (MRI) scoring system that describes tumor mass and is based on 10% increments of the estimated volume of the maximally distended synovial cavity or tendon sheath involved. A tumor that is equal in volume to that of a maximally distended synovial cavity or tendon sheath was scored 10; a score of 0 indicated no evidence of tumor. ORR was the percentage of participants who achieved either CR or PR as assessed by blinded IRR using TVS.
  * CR: Lesion completely gone
  * PR: ≥50% decrease in volume score relative to Baseline.
Time Frame: Baseline to Week 25 (Cycle 7, Day 1)
Population: The ITT Set consisted of participants who were randomized to a study treatment regimen.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vimseltinib | Placebo
Number analyzed (Participants) | 83 | 40
percentage of participants | 67.5 [56.3 to 77.4] | 0 [0.0 to 8.8]
Statistical Analysis 1: Comparison: Vimseltinib vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Stratified by tumor location (lower limb/all other) and region (U.S./non-U.S.) based on IRT; Difference in ORR = 67.2, 95% CI 2-sided [57.0 to 77.3] — Stratified Mantel-Haenszel with stratification factors based on IRT

3. Secondary Outcome: Change From Baseline in Active Range of Motion (ROM) at Week 25
Description: Presented here is the change from baseline in active ROM to Week 25. Measurement of the affected and contralateral, non-affected joint was assessed by goniometer and measured in degrees. At baseline, the motion with the smallest relative ROM value (worst) was identified, and this motion was used for evaluating the change in relative ROM subsequently. The affected joint measurement was used to derive a relative ROM based on active measurement relative to reference standard value provided by the American Medical Association. Relative ROM is expressed in percent: 100 x (joint ROM measure)/(reference ROM standard).
Time Frame: Baseline to Week 25 (Cycle 7, Day 1)
Population: The ITT Set consisted of participants who were randomized to a study treatment regimen. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure at the specified time point.
Measure: Least Squares Mean (Standard Error); unit: Change in percent
Arm/Group | Vimseltinib | Placebo
Number analyzed (Participants) | 73 | 33
Change in percent | 18.4 (6.46) | 3.8 (7.19)
Statistical Analysis 1: Comparison: Vimseltinib vs Placebo; Test type: Superiority; p = 0.0077, Mixed model repeated measures — Model included treatment+visit+treatment by visit interaction+stratification factor for region (U.S. versus non-U.S.)+joint type (knee, ankle, or other)+the most impaired ROM baseline value; LS Mean Difference = 14.6, 95% CI 2-sided [4.0 to 25.3]

4. Secondary Outcome: Change From Baseline in the Patient-reported Outcomes Measurement Information System (PROMIS) Physical Function (PF) Score at Week 25
Description: All participants were asked 15 questions from the PROMIS-PF item bank. The questions used one of two 5-point verbal rating scales: either 1 = "unable to do", 2 = "with much difficulty", 3 = "with some difficulty", 4 = "with a little difficulty", and 5 = "without any difficulty"; or 1 = "cannot do", 2 = "quite a lot", 3 = "somewhat", 4 = "very little", and 5 = "not at all." Total scores were converted to T-scores that ranged from 0 to 100, with higher scores representing less physical function interference and better health outcomes.
Time Frame: Baseline to Week 25 (Cycle 7, Day 1)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vimseltinib | Placebo
Number analyzed (Participants) | 63 | 30
score on a scale | 4.6 (0.96) | 1.3 (0.88)
Statistical Analysis 1: Comparison: Vimseltinib vs Placebo; Test type: Superiority; p = 0.0007, Mixed model repeated measures — Model included treatment+visit+treatment by visit interaction+stratification factor for region (U.S. versus non-U.S.) and tumor location (lower limb/all other) based on IRT+PROMIS-PF baseline value; LS Mean Difference = 3.3, 95% CI 2-sided [1.4 to 5.2]

5. Secondary Outcome: Change From Baseline in the Worst Stiffness Numeric Rating Scale (NRS) Score at Week 25
Description: The Worst Stiffness NRS is a single question that asks the participant to assess their worst stiffness in the last 24 hours. Participants rate their worst stiffness on a scale of 0 to 10, where 0 is "no stiffness" and 10 is "worst imaginable." Lower scores represented better level of stiffness.
Time Frame: Baseline to Week 25 (Cycle 7, Day 1)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vimseltinib | Placebo
Number analyzed (Participants) | 63 | 27
score on a scale | -2.1 (0.24) | -0.3 (0.28)
Statistical Analysis 1: Comparison: Vimseltinib vs Placebo; Test type: Superiority; p < 0.0001, Mixed model repeated measures — Model included treatment+visit+treatment by visit interaction+stratification factor for region (U.S. versus non-U.S.) and tumor location (lower limb/all other) based on IRT+Worst Stiffness NRS baseline value; LS Mean Difference = -1.8, 95% CI 2-sided [-2.5 to -1.1]

6. Secondary Outcome: Change From Baseline in EuroQoL Visual Analogue Scale (EQ-VAS) at Week 25
Description: The EQ-VAS is a standardized tool for measuring overall health. EQ-VAS recorded the participant's self-rated health on a vertical VAS scale ranging from a minimum of 0 (worst imaginable health state) to a maximum of 100 (best imaginable health state). Higher scores indicated better health state.
Time Frame: Baseline to Week 25 (Cycle 7, Day 1)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Vimseltinib | Placebo
Number analyzed (Participants) | 64 | 30
score on a scale | 13.5 (2.35) | 6.1 (2.85)
Statistical Analysis 1: Comparison: Vimseltinib vs Placebo; Test type: Superiority; p = 0.0155, Mixed model repeated measures — Model included treatment+visit+treatment by visit interaction+stratification factor for region (U.S. versus non-U.S.) and tumor location (lower limb/all other) based on IRT+VAS baseline value; LS Mean Difference = 7.4, 95% CI 2-sided [1.4 to 13.4]

7. Secondary Outcome: Percentage of Participants With Response at Week 25 Based on Brief Pain Inventory (BPI) Worst Pain NRS Score and Narcotic Analgesic Use
Description: Participants reported responses to the BPI Worst Pain NRS. The BPI Worst Pain NRS ranged from 0 to 10, where 0 is "no pain" and 10 is "pain as bad as you can imagine." A responder was defined as a participant who:
  (i) experienced a decrease of at least 30% in the mean BPI Worst Pain NRS item and (ii) did not experience a 30% or greater increase in narcotic analgesic use.
Time Frame: Baseline to Week 25 (Cycle 7, Day 1)
Population: The ITT Set consisted of participants who were randomized to a study treatment regimen.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Vimseltinib | Placebo
Number analyzed (Participants) | 83 | 40
percentage of participants | 48.2 [37.1 to 59.4] | 22.5 [10.8 to 38.5]
Statistical Analysis 1: Comparison: Vimseltinib vs Placebo; Test type: Superiority; p = 0.0056, Cochran-Mantel-Haenszel — Stratified by tumor location (lower limb/all other) and region (U.S./non-U.S.) based on IRT; Difference in responder rate = 26.2, 95% CI 2-sided [9.5 to 42.8] — Stratified Mantel-Haenszel with stratification factors based on IRT

ADVERSE EVENTS:
Time Frame: Collection of adverse events started from the signing of informed consent through safety follow-up (up to 1.68 years)
Groups:
- Total - Vimseltinib: Participants received blinded treatment of vimseltinib 30 mg BIW for 24 weeks in Part 1 and/or open-label vimseltinib 30 mg BIW in Part 2 until EoT.
- Placebo: Participants received blinded treatment of matching placebo BIW for 24 weeks.
Arm/Group | Total - Vimseltinib | Placebo
All-Cause Mortality (participants affected / at risk) | 1/118 | 0/39
Serious Adverse Events (participants affected / at risk) | 17/118 | 1/39
Other Adverse Events (participants affected / at risk) | 113/118 | 32/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total - Vimseltinib (N=118) | Placebo (N=39)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 4 (5) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 1 (1) | 0 (0)
Rhinovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total - Vimseltinib (N=118) | Placebo (N=39)
Anaemia (Blood and lymphatic system disorders) | 6 (11) | 2 (2)
Dry eye (Eye disorders) | 9 (9) | 0 (0)
Eyelid oedema (Eye disorders) | 11 (19) | 2 (2)
Lacrimation increased (Eye disorders) | 10 (12) | 0 (0)
Periorbital oedema (Eye disorders) | 53 (87) | 5 (6)
Vision blurred (Eye disorders) | 7 (7) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 3 (4)
Constipation (Gastrointestinal disorders) | 6 (7) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 18 (20) | 7 (8)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 26 (33) | 8 (9)
Vomiting (Gastrointestinal disorders) | 11 (13) | 1 (1)
Asthenia (General disorders) | 30 (51) | 9 (10)
Face oedema (General disorders) | 34 (61) | 3 (3)
Fatigue (General disorders) | 31 (46) | 6 (6)
Generalised oedema (General disorders) | 16 (32) | 0 (0)
Oedema peripheral (General disorders) | 20 (29) | 3 (3)
Pyrexia (General disorders) | 8 (12) | 0 (0)
COVID-19 (Infections and infestations) | 16 (16) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 17 (19) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 30 (47) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 26 (82) | 0 (0)
Blood creatinine increased (Investigations) | 7 (12) | 1 (1)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 7 (10) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 7 (10) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 (38) | 6 (7)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (14) | 3 (4)
Dizziness (Nervous system disorders) | 6 (6) | 2 (3)
Headache (Nervous system disorders) | 30 (49) | 10 (16)
Paraesthesia (Nervous system disorders) | 10 (17) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3) | 2 (2)
Insomnia (Psychiatric disorders) | 8 (9) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 10 (12) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 9 (9) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 33 (52) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 25 (44) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 22 (31) | 0 (0)
Hypertension (Vascular disorders) | 18 (34) | 4 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-05-31): https://cdn.clinicaltrials.gov/large-docs/62/NCT05059262/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT05059262/SAP_001.pdf